CLINICAL TRIAL: NCT06122571
Title: A Clinical Trial to Evaluate the Effect of ConcenTrace Trace Mineral Drops on Gut Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trace Minerals (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20351
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Gut Health; Bowel Movements; Constipation; Bloating
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test arm: ConcenTrace (Experimental): Participants will follow this weekly dosing schedule:
  Week 1: Day 1-3: take 5 drops of ConcenTrace with 8oz of water or flavored water. Day 4-7: take 5 drops of ConcenTrace 2x per day with 8 oz of water or flavored water.
  Week 2: Take 10 drops of ConcenTrace 2x per day with 8 oz of water or flavored water.
  Week 3: Take 15 drops of ConcenTrace 2x per day with 8 oz of water or flavored water.
  Week 4: Take 20 drops of ConcenTrace 2x per day with 8 oz of water or flavored water.
  Weeks 5 - 12: Take 40 drops of ConcenTrace 1x per day with 8 oz of water or flavored water.
  Interventions: Other: ConcenTrace

INTERVENTIONS:
Other: ConcenTrace — The product contains concentrated seawater from Utah's inland sea.

SUMMARY:
This is a virtual single-arm trial that will last 12 weeks. Participants will take the drops daily and complete questionnaires at Baseline, Week 4, Week 8, and Week 12. Gut health, bowel movements, stool looseness, constipation, bloating, and regularity will be evaluated at the Baseline and at each check-in. Likert scale responses will be statistically compared from Baseline to each check-in. Participant responses and product feedback will be presented as percentage scores.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female. Be aged over 18. Have a BMI less than 35. Have issues with digestion, heartburn, indigestion, gas, or constipation. Be willing to maintain their standard dietary pattern, activity level, and body weight for the duration of the study.

Be generally healthy - must not live with any uncontrolled disease.

Exclusion Criteria:

* Any person with a pre-existing chronic condition that might prevent the participant from adhering to the protocol, including any oncological and psychiatric disorders.

Anyone taking any prescribed medication targeting the gut. Anyone taking any supplements targeting the gut within the past month. Anyone with any known severe allergic reactions. Women who are pregnant, breastfeeding, or attempting to become pregnant. Anyone unwilling to follow the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in scores on the Gastrointestinal Symptom Rating Scale (GSRS). [Timeframe: Baseline to Week 12] | 12 weeks
  The GSRS is a disease-specific instrument of 15 items combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.

SECONDARY OUTCOMES:
Changes in stool consistency reported via the Bristol Stool Chart. [Timeframe: Baseline to Week 12] | 12 weeks
  The Bristol stool scale is a diagnostic medical tool designed to classify the form of human faeces into seven categories. Type 1 has spent the longest time in the bowel and type 7 the least time.
Changes in bowel movement frequency. [Timeframe: Baseline to Week 12] | 12 weeks
  The frequency that the participants have a bowel movement will be recorded via questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided